CLINICAL TRIAL: NCT05614388
Title: A Study on Utilization, Adherence, and Acceptability of Voluntary Routine COVID-19 Self-testing Among Students, Staff and Health Workers at Two Institutions in Mizoram, India.
Brief Title: A Study on Voluntary Routine COVID-19 Self-testing in Mizoram, India.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PATH (Other)
Collaborators: UNITAID (Other); Zoram Medical College (ZMC) (Unknown); Pacchunga University College (Unknown); Association for Leprosy Education Rehabilitation & Treatment India (ALERT India) (Unknown); Government of Mizoram (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RES-376
Record Dates: First submitted 2022-11-09; First posted 2022-11-14 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: COVID 19; Self-Test; Pandemic Preparedness; Infectious diseases
MeSH Terms: conditions — COVID-19; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: The participants include health care workers, non-medical hospital staff and medical students at ZMC; and faculty, students and supporting staff at the Pacchunga University College. All these groups will be participating in the study simultaneously. The study results will be compared for all these 6 groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): The study procedure is universal to all the participants from both the institutes. There are no control arms defined separately. The groups within the participants include - include health care workers, non-medical hospital staff and medical students at ZMC; and faculty, students and supporting staff at the Pacchunga University College.
  Interventions: Diagnostic Test: COVID-19 Self testing and related messaging

INTERVENTIONS:
Diagnostic Test: COVID-19 Self testing and related messaging — Provisioning of voluntary, free self-testing for COVID-19 (approved and validated in the country) and related Information, Education and Communication (IEC) messages

SUMMARY:
This interventional study aims to evaluate the utilization, adherence, and acceptability of voluntary, free, routine self-testing for COVID-19 (Corona Virus (19) Disease) and related information, education and communication (IEC) messages in two institutional settings in Mizoram, India. In addition, it will assess and measure preferences for assisted vs unassisted and observed vs unobserved self-testing, assess adherence and measure dropout rate and describe dropout characteristics.

The research questions it aims to address are -

1. What is the uptake and adherence of voluntary, free, routine self-testing for COVID-19 and related IEC messages vy students, employees, and healthcare workers in two institutional settings in India? Are there any dropouts from routine self-testing and what are the factors related to dropouts?
2. What is the preferred mode of self-testing- observed or unobserved, assisted or unassisted? Do these preferences change over time? The researchers will be measuring - Utilization rate, Adherence rate, Proportion of preference to assisted vs unassisted self-testing, Proportion of preference to observed vs unobserved self-testing, Time to dropout and Acceptability of COVID-19 self-testing kits.

DETAILED DESCRIPTION:
Testing is a critical component of the pandemic response. It serves two purposes; for clinical purposes, it focuses on identifying disease in symptomatic patients, while testing for epidemiological purposes, spread in the population is also assessed. India uses a mix of both Reverse Transcriptase Polymerase Chain Reaction (RT PCR) and Antigen Rapid Diagnostic Tests (Ag RDTs) for COVID-19 testing. RT PCR is the reference standard test for detection of the virus. However, not all facilities have RT PCR, and many communities have poor access. This leads to a long turn-around time (TAT) for the results to be obtained and a high load on RT PCR facilities. Hence, to prevent the spread of the virus, cases must get detected early. At the peak of the first wave of the pandemic in the country, Ag RDTs constituted close to 50% of all the tests conducted in the country. Self-testing for COVID-19 has emerged as a viable complementary testing modality. The use of self-testing kits while ensuring the availability of other COVID-19 tests at the nearest point of care addresses many of the usual barriers to uptake of services, leading to timely testing of individuals, diagnosis, and access to care. It can also reduce the burden on existing testing infrastructure especially during a surge in the cases. It also reduces overcrowding at testing facilities thereby reducing the risk of disease transmission. To improve access to testing and prevent overreliance on RT PCR laboratories, the Indian Council of Medical Research (ICMR) approved and validated the use of COVID-19 self-testing kits. As of March 2022, sixteen self-testing kits have been validated in India of which 10 are found to be satisfactory. While there are many benefits to self-testing, it is also essential to understand the utilization of the self-testing strategy, including whether or not the community can follow the steps for self-testing and what support, if any, the community may require to use self-test kits.

The present study proposes the demonstration of ICMR and US-FDA (United States Food & Drug Administration) approved SURE STATUS self-testing kit in the healthcare workers and educational institution setting in Mizoram for a period of 5 months. With the ease of lockdown and movement restrictions, workplaces and educational institutes are gradually opening up. However, with the threat of the pandemic still looming large, it is prudent to put in place systems for regular screening within these settings to promote early diagnosis and care and prevent outbreaks. COVID-19 self-test has been identified as one way any institution can scale up COVID-19 testing to improve COVID-19 status awareness by reaching out to as many people as possible at a given point of time.

While COVID-19 self-tests are available and widely used in India, these kits are largely used within the confines of individual homes. It is learnt that the reporting of the results of the self-test is poor as compared to the utilization of the self-test kits. To the investigator's knowledge, no study has been conducted in India to assess the utilization of self-testing as a routine procedure in places of mass indoor gathering, like workplaces and educational institutions. To address this gap, the investigators will conduct a study to evaluate the utilization, adherence, and acceptability of routine COVID-19 self-testing among students, employees and healthcare workers in two congregate settings: one University College and one Medical College and Hospital in Mizoram, India. The proposed study will document challenges, if any, in reporting of self-test results and document the key processes in operationalizing routine COVID-19 self-testing among students, employees and healthcare workers and provide learning and recommendations for systematic use of self-tests for future models of institution based COVID-19 self-testing in congregate settings.

ELIGIBILITY:
Inclusion Criteria:

1. Above the age of 18 years, irrespective of gender and past COVID-19 status
2. Registered with participating institutions
3. Able and willing to provide informed consent
4. Owns a smartphone capable of downloading the SURE STATUS app for uploading results
5. Able to read the instructions in the Mizo or English or Hindi

Exclusion Criteria:

1. Does not consent.
2. Has any contraindication to nasal sample collection, including recent nasal injury, nasal surgeries.
3. Personnel who are directly involved in the conduct of the study, e.g., investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 646 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Utilization rate | 5 Months
  Individual level: the proportion of tests each individual uses till the end of the follow-up period from the minimum number of tests allocated to them.
  Sample-level: mean and standard deviations calculated based on the individual utilisation rates
Adherence Rate | 5 Months
  Individual level: the proportion of tests an individual performs according to the testing schedule over the total number of tests they perform.
  Sample-level: mean and standard deviations calculated based on the individual adherence rates
Preferences of participants on self testing | 5 Months
  Proportion of preference to assisted vs unassisted self-testing
Observation proportions of participants on self testing | 5 Months
  Proportion of preference to observed vs unobserved self-testing
Time to dropout | 5 Months
  The time to drop out will be the time from enrolment of the participant till drop-out
Acceptability of COVID-19 self-testing kits | 5 Months
  A composite indicator based on ease of use of COVID-19 self-testing kits, ease of interpretation of test results, and recommendation to others

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ralte, MD, Principal Investigator — Zoram Medical College

IPD SHARING:
Plan to Share IPD: No
We do not plan to share any individual participant data. We will share collective learnings on various parameters at both the sites.